CLINICAL TRIAL: NCT00935194
Title: Antiviral and Chinese Medicinal Herbs Treatment on Novel Influenza A (H1N1) Virus Infection: Multi-centre, Prospective, Randomized Controlled Study
Brief Title: Chinese Medicinal Herbs Treatment on Novel Influenza A (H1N1) : Multi-centre, Prospective, Randomized Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Wang Chen, Capital Medical University Affiliated Beijing Chaoyang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z09000700090903
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Influenza
Keywords: Novel Influenza A(H1N1); Oseltamivir; Chinese Medicinal Herbs
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- blank (Experimental): do not take antiviral therapy
  Interventions: Other: blank
- Oseltamivir (Experimental): antiviral therapy
  Interventions: Drug: oseltamivir
- chinese medicinary herbs (Experimental): antiviral therapy
  Interventions: Drug: chinese medicinal herbs
- oseltalmivir and chinese medicinal herbs (Experimental): combination antiviral therapy
  Interventions: Drug: oseltamivir and chinese medicinal herbs

INTERVENTIONS:
Drug: oseltamivir — 75mg,bid,for 5 days
  Other Names: TamifluTM
  Arms: Oseltamivir
Other: blank — no antiviral therapy
  Arms: blank
Drug: chinese medicinal herbs — 200ml,p.o,qid,for 5 days
  Arms: chinese medicinary herbs
Drug: oseltamivir and chinese medicinal herbs — oseltamivir:75mg,p.o,bid,for 5 days; chinese medicinal herbs:200ml,p.o,qid,for 5 days
  Arms: oseltalmivir and chinese medicinal herbs

SUMMARY:
The purpose of this study is to determine whether Chinese medicinal herbs are effective and safe for treating novel influenza A (H1N1) infection.

DETAILED DESCRIPTION:
The antiviral agent, oseltamivir, is recommended by the World Health Organization (WHO) to treat recent outbreak novel influenza A (H1N1) virus infection around world. But limited stock and resistant strain emergence raised increasing concerns. Chinese medicinal herbs, are derived from plants and usually incorporate one or more herbs as the basic drug(s) to treat the disease. The investigators performed RCT to indicate that Chinese medicinal herbs was effective and safe for treating novel influenza A (H1N1) infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed novel influenza A(H1N1) case with laboratory evidence
* 70 years ≥ age ≥ 14years
* Within 72hr after the onset of symptoms(body temperature≥37.5℃ with at least one respiratory symptom (cough, sore throat, or nasal symptom)

Exclusion Criteria:

* Age < 14 years or > 70 years
* Bronchitis, pneumonia, pleural fluid and interstitial infiltration showed by Chest radiology(x-ray or CT)
* Severe chronic underlying diseases: severe COPD(FEV1/EVC <70% and FEV1 <30% predicted or respiratory failure or congestive heart failure), severe hepatic disfunction（ALT or AST ≥3 times normal elevation), renal disfunction（Cr>2mg/dL), chronic heart failure(NYHA Ⅲ-Ⅳ grade）
* Immunocompromised patients(cancer, organ transplant, AIDS and a history of treatment with immunosuppressive drug and glucocorticoids in the past 3 months)
* Taken Chinese medicinal herbs, antiviral or antibiotic drug in the past 2 weeks
* Inoculation influenza vaccination
* One of the following items appeared at the enrollment

  * respiratory failure：PaO2<60mmHg and/or PCO2>50mmHg or PaO2/FiO2≤300
  * circulation failure: despite adequate fluid resuscitation and cardiac output, systolic <90mmHg or requirement inotropic support
  * renal function failure: despite adequate fluid resuscitation and cardiac output, urine ≤ 0.5ml/kg.h, Cr or BUN≥1 time normal elevation
  * hepatic function failure: total bilirubin>34μmol/L or ALT/AST ≥3 times normal - Other unappropriated enrollment situations considered by investigator

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
time to resolution of fever (the period from start of study-drug to relief of fever) | one year

SECONDARY OUTCOMES:
time to resolution of respiratory symptoms(defined as the period from start of study-drug to relief of symptoms) | one year
virus shedding time | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Doctor, Study Chair — Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute; Qingquan Liu, Docter, Principal Investigator — Beijing Chinese Traditional Medicine University affiliated Dongzhimen Hospital; Yu Mao, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute, Beijing, China

REFERENCES:
- [Derived] Wang C, Cao B, Liu QQ, Zou ZQ, Liang ZA, Gu L, Dong JP, Liang LR, Li XW, Hu K, He XS, Sun YH, An Y, Yang T, Cao ZX, Guo YM, Wen XM, Wang YG, Liu YL, Jiang LD. Oseltamivir compared with the Chinese traditional therapy maxingshigan-yinqiaosan in the treatment of H1N1 influenza: a randomized trial. Ann Intern Med. 2011 Aug 16;155(4):217-25. doi: 10.7326/0003-4819-155-4-201108160-00005. PMID 21844547